CLINICAL TRIAL: NCT01937234
Title: Use of an Antiemetic to Shorten the Length of Labor in Nulliparous Women, Exploring a Potential Role of an Old Drug
Brief Title: Use of an Antiemetic to Shorten the Length of Labor in Nulliparous Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Lecturer of Obstetrics & Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AFHSR-13-7-2013
Record Dates: First submitted 2013-09-01; First posted 2013-09-09 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Prolonged First Stage of Labor
MeSH Terms: interventions — Metoclopramide; Patents as Topic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoclopramide (Active Comparator): Intravenous injection of 10mg metoclopramide
  Interventions: Drug: Metoclopramide
- Placebo (Placebo Comparator): Intravenous injection of 0.9% sodium chloride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide — Intravenous injection of 10mg metoclopramide, at enrollment, then every 2 hours.
  Maximum of 3 doses.
  Other Names: Primperan (Trademark)
  Arms: Metoclopramide
Drug: Placebo — Intravenous injection of 0.9% sodium chloride, at enrollment, then every 2 hours.
  Maximum of 3 doses.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Reducing the length of labor is a highly desirable goal of intrapartum care, both from a perspective of maternal and fetal well-being , and for the providers of the birth services. Avoiding a long , protracted labor entails shorter exposure to pain anxiety and stress and would translate into a major improvement in maternal satisfaction with the child birth experience.

The purpose of this study is to determine the effectiveness of metoclopramide for reducing the duration of spontaneous labor among nulliparous women managed according to a standard intrapartum protocol.

DETAILED DESCRIPTION:
Women who will fulfill the study inclusion and exclusion criteria and agree to be included in the study will be randomized assigned to receive either an intravenous injection of 10mg metoclopramide (Group 1) or the same volume of placebo, i.e. 0.9% sodium chloride (Group2). Randomization will be achieved using computer generated randomization sequences. Allocation will be in 1:1 ratio. Record of group allocation will be maintained by a resident physician whose responsibility is randomization and drawing up the injection, but has no direct involvement in the intrapartum decision making.

After through history and physical examination, each participant will take the selected medication slowly IV over 2 min, the assigned medication will be repeated every two hours for a maximum of three doses.

Monitoring of fetal well-being and labor progress with Partographic representation will be performed.

Management of labor will be according the labor and delivery standard protocol, if labor dilatation will not progress appropriately, i.e. cervical dilatation rate of <1cm/hour, amniotomy will be performed if membranes are intact. Oxytocin augmentation will be considered after rupture of membranes only if the cervix remains unchanged on two consecutive pelvic examination conducted two hours apart. Oxytocin infusion will start with 5mIU/min and increase by 5mIU/min every 15min to achieve seven contractions in 15 min, the maximal rate of oxytocin being 30Miu/min.

The following parameters will be recorded for every patient:

* Timing of metoclopramide or placebo injections
* Timing of full dilatation of cervix
* Duration of first stage of labor
* Duration of second stage of labor
* Duration of third stage of labor
* Mode of delivery
* Injection to delivery interval
* Cervical dilatation rate
* Neonatal condition at birth

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* Singleton pregnancy
* Term gestation i.e. 37- 42 weeks
* Sure reliable dates
* Vertex presentation, occipitoanterior position
* Spontaneous onset of labor
* Regular uterine contractions at every 5 min ,each lasting for 20 sec
* Cervical dilatation of 3-5cm
* With or without rupture of membranes
* No evidence of maternal or fetal distress

Exclusion Criteria:

* Mal-presentations
* Mal-positions
* Multifetal pregnancy
* Cephalopelvic disproportion
* history of cervical surgery or injury
* Hypersensitivity to metoclopramide

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cervical dilatation rate | 6 hours

SECONDARY OUTCOMES:
Duration of the first stage of labor | 6 hours

OTHER OUTCOMES:
Duration of the second stage of labor | 2 hours
Duration of the third stage of labor | 1 hour
Number of Participants with Adverse Events | 24 hours
  Adverse effects of metoclopramide:
  * Cardiovascular: heart block, bradycardia, heart failure, flushing, hyper or hypotension, supraventricular tachycardia.
  * Central nervous system: Drowsiness, acute dystonic reactions, headache, dizziness, akathisia, confusion, depression, hallucinations, Parkinsonian-like symptoms, suicidal ideation, seizure, tardive dyskinesia
  * Dermatologic: Angioneurotic edema, rash, urticaria
  * Gastrointestinal: Nausea, vomiting, diarrhea
  * Respiratory: Bronchospasm, laryngeal edema (rare), laryngospasm (rare)
Apgar score | 10 minutes
Meconium stained liquor | 6 hours
Neonatal intensive care unit admission rate | 24 hours
Rate of vaginal delivery | 12 hours
Number of participants with genital tract injuries | 2 hours
  genital tract injuries:
  * Perineal tears
  * Vaginal tears
  * Cervical tears
  * Perineal hematomas
  * Vaginal hematomas
  * Uterine rupture

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Ellaithy, MD, Study Director — Ain Shams University
Locations (1):
- Labor and delivery ward of Armed Forces Hospital, Southern Region., Khamis Mushait, Khamis Mushait, Saudi Arabia

REFERENCES:
- [Derived] Ellaithy M, Rasheed S, Shafik A, Abees S. Use of an antiemetic to shorten the length of labor in nulliparous women, exploring a potential role of an old drug: A randomized controlled trial. Int J Gynaecol Obstet. 2020 Jan;148(1):72-78. doi: 10.1002/ijgo.12998. Epub 2019 Nov 8. PMID 31609464